CLINICAL TRIAL: NCT04872049
Title: Assessment of SARS-CoV-2 Effect on Post-traumatic Stress of Patients Hospitalized in Intensive Care
Brief Title: Assessment of SARS-CoV-2 Effect on Post-traumatic Stress of Patients Hospitalized in Intensive Care Unit
Acronym: FAMILY-COVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200450; 2020-A03430-39 (Other: IDRCB)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Intensive Care Unit; SARS-CoV2
Keywords: SARS-CoV-2; Post-traumatic stress; Anxiety; Depression; Covid-19; Intensive-care
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients admitted to the intensive care unit develop psychiatric disorders, such as anxiety, depression or post-traumatic stress disorder, which can be prolonged.

During the COVID crisis, the presence of relatives in the intensive care unit was reduced and this, in a lasting way.

The hypothesis is that there is a difference in the experience of the stay in the intensive care unit whether or not one is affected by SARS-CoV-2 and that this difference is likely to have an impact on the long-term outcome of the patients and their relatives.

DETAILED DESCRIPTION:
The stay in the ICU is a complex and often traumatic experience for patients. Patients often develop psychiatric disorders such as anxiety, depression or post-traumatic stress disorder after an ICU stay. These symptoms can be prolonged over time, resulting in a decrease in quality of life and a potential cost in care.

In the epidemic context of the COVID crisis, the presence of family members in the intensive care unit was reduced to its most extreme portion, with sometimes an almost total impossibility of visiting a loved one. This situation, although it has become less strict, has lasted for a long time. The patient can only exchange with them with difficulty, despite the extremely trying situation that is resuscitation. Moreover, there is a stress factor linked to the infectious risk for the relatives and for the relatives with regard to COVID-19, in particular within the framework of family clusters with sometimes several hospitalized subjects within the same family.

Of course, means of communication have been put in place with relatives, but these means do not seem to be equivalent to the presence of one's relatives.

The investigators therefore hypothesize that there is a difference in the experience of the stay in the intensive care unit whether or not one is affected by SARS-CoV-2 and that this difference is likely to have an impact on the long-term outcome of patients and their relatives.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (above 18 years old)
* Admitted in intensive care unit
* Hospitalized more than 2 days (48 hours)
* Between 01/01/2020 and 06/30/2020
* Whether SARS-CoV-2 positive or negative

Exclusion Criteria:

* Minor patient
* Protected major (under safeguardship, curatorship or guardianship)
* Patient opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted more than 2 days (48 hours) in Intensive care unit between 01/01/2020 and 06/30/2020i, infected or not with SARS-CoV-2;
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-10-27 (Estimated); Study Completion 2021-10-27 (Estimated)

PRIMARY OUTCOMES:
Prevalence of post-traumatic stress at 1 year | 12 months from hospitalization
  Prevalence of post-traumatic stress in patients treated in intensive care at 1 year diagnosed with an IES-r> 33 depending on whether they are SARS-CoV-2 positive or not.
  (IES-r: Impact of Event Scale - Revised scale, minimum value: 0, maximum value: 88, higher score indicates a worse outcome)

SECONDARY OUTCOMES:
Level of depression at 1 year | 12 months from hospitalization
  Assessed by the Center for Epidemiologic Studies Depression scale (CES-D, minimum value: 0, maximum value: 60, higher score indicates a worse outcome)
Perceived interest of the proposed communication tools at 1 year | 12 months from hospitalization
  Semi-structured interviews
Level of quality of life at 1 year | 12 months from hospitalization
  Assessed by EQ-5D (EuroQol 5Dimension scale, minimum value: 0, maximum value: 100, higher score indicates a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Claire FAZILLEAU, Study Director — Assistance Publique - Hôpitaux de Paris; Arthur Dr JAMES, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- GH Pitié Salpêtrière - Charles Foix, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No